CLINICAL TRIAL: NCT03070899
Title: A Phase 3, Multicentre, Randomized, Double-blind, Placebo-controlled Study Investigating the Efficacy and Safety of Daily Oral Administration of OBE2109 Alone and in Combination With Add-back Therapy for the Management of Heavy Menstrual Bleeding Associated With Uterine Fibroids in Premenopausal Women
Brief Title: Efficacy and Safety of OBE2109 in Subjects With Heavy Menstrual Bleeding Associated With Uterine Fibroids
Acronym: PRIMROSE 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ObsEva SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-OBE2109-008
Record Dates: First submitted 2017-02-17; First posted 2017-03-06 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Uterine Fibroids; Heavy Menstrual Bleeding
Keywords: Uterine Fibroid; Leiomyomata; Heavy Menstrual Bleeding; HMB; Heavy Uterine Bleeding; Menorrhagia; OBE2109 + Add-back
MeSH Terms: conditions — Leiomyoma; Menorrhagia | interventions — linzagolix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- OBE2109 dose 1 (100mg) + Placebo Add-back (Experimental)
  Interventions: Drug: OBE2109; Drug: Placebo to match OBE2109; Drug: Placebo to match Add-back
- OBE2109 dose 1 (100mg) + Add-back (Experimental)
  Interventions: Drug: OBE2109; Drug: Placebo to match OBE2109; Drug: Add-back
- OBE2109 dose 2 (200mg) + Placebo Add-back / OBE2109 dose 2 (200 mg) + Add-back (Experimental)
  Interventions: Drug: OBE2109; Drug: Placebo to match Add-back; Drug: Add-back
- OBE2109 dose 2 (200mg) + Add-back (Experimental)
  Interventions: Drug: OBE2109; Drug: Add-back
- Placebo + Placebo Add-back / OBE2109 dose 3 (200mg) + Add-back (Placebo Comparator): At W24, half of the patients switched to active treatment, while half remained on Placebo; the switch was defined at randomization.
  Interventions: Drug: OBE2109; Drug: Placebo to match OBE2109; Drug: Placebo to match Add-back; Drug: Add-back

INTERVENTIONS:
Drug: OBE2109 — OBE2109 100mg tablets for oral administration once daily
Drug: Placebo to match OBE2109 — Placebo to match OBE2109 100mg tablets for oral administration once daily
  Arms: OBE2109 dose 1 (100mg) + Add-back; OBE2109 dose 1 (100mg) + Placebo Add-back; Placebo + Placebo Add-back / OBE2109 dose 3 (200mg) + Add-back
Drug: Placebo to match Add-back — Placebo to match Add-back (E2 1 mg / NETA 0.5 mg) for oral administration once daily
  Arms: OBE2109 dose 1 (100mg) + Placebo Add-back; OBE2109 dose 2 (200mg) + Placebo Add-back / OBE2109 dose 2 (200 mg) + Add-back; Placebo + Placebo Add-back / OBE2109 dose 3 (200mg) + Add-back
Drug: Add-back — Add-back (E2 1 mg / NETA 0.5 mg) for oral administration once daily
  Arms: OBE2109 dose 1 (100mg) + Add-back; OBE2109 dose 2 (200mg) + Add-back; OBE2109 dose 2 (200mg) + Placebo Add-back / OBE2109 dose 2 (200 mg) + Add-back; Placebo + Placebo Add-back / OBE2109 dose 3 (200mg) + Add-back

SUMMARY:
The primary objective of this study is to demonstrate the superior efficacy versus placebo of OBE2109 alone and in combination with add-back therapy for the reduction of heavy menstrual bleeding associated with uterine fibroids in premenopausal women.

DETAILED DESCRIPTION:
The study is a prospective, randomized, parallel group, double-blind, placebo-controlled phase 3 study investigating the efficacy and safety of OBE2109 alone and in combination with add-back therapy for the treatment of uterine fibroids.

Subjects will be randomized to one of 5 treatment groups in a 1:1:1:1:1 ratio.

ELIGIBILITY:
Key Inclusion Criteria:

* Premenopausal woman at screening.
* Body Mass Index ≥ 18 kg/m2.
* Menstrual cycles ≥ 21 days and ≤ 40 days.
* Presence of uterine fibroids.
* Heavy menstrual blood loss for each of the 2 menstrual periods assessed at screening using the alkaline hematin method.

Key Exclusion Criteria:

* The subject is pregnant or breast-feeding or is planning a pregnancy within the duration of the treatment period of the study.
* History of uterus surgery that would interfere with the study.
* The subject's condition is so severe that she will require surgery within 6 months regardless of the treatment provided.
* Undiagnosed abnormal uterine bleeding.
* Significant risk of osteoporosis or history of, or known osteoporosis or other metabolic bone disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
Percentage of Responders based on menstrual blood loss (MBL) volume reduction at Week 24 | From baseline to Week 24
  Assessed using the alkaline hematin method

SECONDARY OUTCOMES:
Time to reduced menstrual blood loss | Up to Week 52
  Assessed using the alkaline hematin method
Amenorrhea | Up to Week 52
  Assessed using the alkaline hematin method
Time to amenorrhea | Up to Week 52
Number of days of uterine bleeding for the last 28-day interval prior to Week 24 | last 28-day interval prior to Week 24
  Assessed using the alkaline hematin method
Number of days of uterine bleeding for each 28-day interval | Up to Week 52
  Assessed using the alkaline hematin method

OTHER OUTCOMES:
Bone Mineral Density (BMD) | From baseline up to Week 76
  Assessed by dual-energy X-ray absorptiometry (DXA) scan
Endometrial biopsy | From baseline up to Week 52
  Assessed by histology
Adverse events | Up to Week 76
  Frequency and severity of Treatment-Emergent Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: ObsEva SA, Study Director — Geneva
Locations (116):
- United States (116):
  - Site reference ID 192, Birmingham, Alabama
  - Site reference ID 169, Dothan, Alabama
  - Site reference ID 353, Mobile, Alabama
  - Site reference ID 232, Vestavia Hills, Alabama
  - Site reference ID 242, Phoenix, Arizona
  - Site reference ID 355, Tucson, Arizona
  - Site reference ID 211, Arcadia, California
  - Site reference ID 184, Cerritos, California
  - Site reference ID 147, Escondido, California
  - Site reference ID 154, Huntington Park, California
  - Site reference ID 185, Los Angeles, California
  - Site reference ID 199, Northridge, California
  - Site reference ID 111, Panorama City, California
  - Site reference ID 166, Sacramento, California
  - Site reference ID 101, San Diego, California
  - Site reference ID 239, Upland, California
  - Site reference ID 112, Westminster, California
  - Site reference ID 144, Denver, Colorado
  - Site reference ID 246, Englewood, Colorado
  - Site reference ID 234, Thornton, Colorado
  - Site reference ID 189, New Haven, Connecticut
  - Site reference ID 105, Washington D.C., District of Columbia
  - Site reference ID 231, Boca Raton, Florida
  - Site reference ID 190, Boca Raton, Florida
  - Site reference ID 168, Clearwater, Florida
  - Site reference ID 233, DeLand, Florida
  - Site reference ID 197, Fort Lauderdale, Florida
  - Site reference ID 135, Hialeah, Florida
  - Site reference ID 146, Hialeah, Florida
  - Site reference ID 191, Jacksonville, Florida
  - Site reference ID 204, Loxahatchee Groves, Florida
  - Site reference ID 137, Miami, Florida
  - Site reference ID 142, Miami, Florida
  - Site reference ID 110, Miami, Florida
  - Site reference ID 106, Miami, Florida
  - Site reference ID 127, Miami, Florida
  - Site reference ID 117, Miami Lakes, Florida
  - Site reference ID 134, Miami Lakes, Florida
  - Site reference ID 129, Miami Springs, Florida
  - Site reference ID 107, Miramar, Florida
  - Site reference ID 124, New Port Richey, Florida
  - Site reference ID 141, Orlando, Florida
  - Site reference ID 140, Orlando, Florida
  - Site reference ID 207, St. Petersburg, Florida
  - Site reference ID 113, Tampa, Florida
  - Site reference ID 163, Columbus, Georgia
  - Site reference ID 158, Norcross, Georgia
  - Site reference ID 151, Norcross, Georgia
  - Site reference ID 150, Sandy Springs, Georgia
  - Site reference ID 359, Idaho Falls, Idaho
  - Site reference ID 352, Meridian, Idaho
  - Site reference ID 174, Champaign, Illinois
  - Site reference ID 182, Oak Brook, Illinois
  - Site reference ID 178, Shawnee Mission, Kansas
  - Site reference ID 354, Wichita, Kansas
  - Site reference ID 176, Lake Charles, Louisiana
  - Site reference ID 109, Marrero, Louisiana
  - Site reference ID 248, Frederick, Maryland
  - Site reference ID 226, Silver Spring, Maryland
  - Site reference ID 228, Towson, Maryland
  - Site reference ID 149, Fall River, Massachusetts
  - Site reference ID 126, Fall River, Massachusetts
  - Site reference ID 100, Bay City, Michigan
  - Site reference ID 145, Detroit, Michigan
  - Site reference ID 214, Saginaw, Michigan
  - Site reference ID 170, Saginaw, Michigan
  - Site reference ID 138, Missoula, Montana
  - Site reference ID 236, Las Vegas, Nevada
  - Site reference ID 245, Lawrenceville, New Jersey
  - Site reference ID 175, Brooklyn, New York
  - Site reference ID 188, New York, New York
  - Site reference ID 208, Port Jefferson, New York
  - Site reference ID 133, Staten Island, New York
  - Site reference ID 104, Greensboro, North Carolina
  - Site reference ID 131, Morehead City, North Carolina
  - Site reference ID 102, Raleigh, North Carolina
  - Site reference ID 187, Southern Pines, North Carolina
  - Site reference ID 119, Winston-Salem, North Carolina
  - Site reference ID 186, Cincinnati, Ohio
  - Site reference ID 164, Cleveland, Ohio
  - Site reference ID 230, Fairfield, Ohio
  - Site reference ID 213, Franklin, Ohio
  - Site reference ID 116, Bryn Mawr, Pennsylvania
  - Site reference ID 195, Hershey, Pennsylvania
  - Site reference ID 222, Indiana, Pennsylvania
  - Site reference ID 165, Jenkintown, Pennsylvania
  - Site reference ID 210, Pittsburgh, Pennsylvania
  - Site reference ID 148, Smithfield, Pennsylvania
  - Site reference ID 351, North Charleston, South Carolina
  - Site reference ID 358, Spartanburg, South Carolina
  - Site reference ID 159, Chattanooga, Tennessee
  - Site reference ID 235, Knoxville, Tennessee
  - Site reference ID 205, Memphis, Tennessee
  - Site reference ID 180, Memphis, Tennessee
  - Site reference ID 238, Austin, Texas
  - Site reference ID 155, Austin, Texas
  - Site reference ID 201, Beaumont, Texas
  - Site reference ID 247, Corpus Christi, Texas
  - Site reference ID 183, Dallas, Texas
  - Site reference ID 216, Dallas, Texas
  - Site reference ID 200, Dallas, Texas
  - Site reference ID 250, Fort Worth, Texas
  - Site reference ID 244, Fort Worth, Texas
  - Site reference ID 115, Frisco, Texas
  - Site reference ID 157, Houston, Texas
  - Site reference ID 120, Houston, Texas
  - Site reference ID 219, Houston, Texas
  - Site reference ID 217, Houston, Texas
  - Site reference ID 218, Pasadena, Texas
  - Site reference ID 172, San Antonio, Texas
  - Site reference ID 128, Webster, Texas
  - Site reference ID 125, West Jordan, Utah
  - Site reference ID 103, Norfolk, Virginia
  - Site reference ID 171, Norfolk, Virginia
  - Site reference ID 123, Richmond, Virginia
  - Site reference ID 237, Bellevue, Washington

REFERENCES:
- [Derived] Donnez J, Petraglia F, Taylor H, Becker CM, Becker S, Herrera FC, Bestel E, Hori S, Dolmans MM. Linzagolix with and without hormonal add-back therapy for symptomatic uterine fibroids: PRIMROSE 1 & 2 long-term extension and withdrawal study. Fertil Steril. 2025 Oct;124(4):737-748. doi: 10.1016/j.fertnstert.2025.06.016. Epub 2025 Jun 19. PMID 40543832
- [Derived] Becker S, Dolmans MM, Herrera FC, Petraglia F, Renner SP, Ionescu-Ittu R, St-Pierre J, Boolell M, Bestel E, Hori S, Donnez J. Pain Reduction in Linzagolix-Treated Patients With Uterine Fibroids: A Secondary Mediation Analysis of the PRIMROSE 1 and 2 Phase 3 Trials. BJOG. 2025 Aug;132(9):1297-1306. doi: 10.1111/1471-0528.18190. Epub 2025 May 6. PMID 40326221
- [Derived] Donnez J, Taylor HS, Stewart EA, Bradley L, Marsh E, Archer D, Al-Hendy A, Petraglia F, Watts N, Gotteland JP, Bestel E, Terrill P, Loumaye E, Humberstone A, Garner E. Linzagolix with and without hormonal add-back therapy for the treatment of symptomatic uterine fibroids: two randomised, placebo-controlled, phase 3 trials. Lancet. 2022 Sep 17;400(10356):896-907. doi: 10.1016/S0140-6736(22)01475-1. PMID 36116480